CLINICAL TRIAL: NCT03141879
Title: Assessing the Feasibility and Impact of an Adapted Resistance Training Intervention, Aimed at Improving the Multi-dimensional Health and Functional Capacity of Frail Older Adults in Residential Care Settings: Protocol for a Feasibility Study
Brief Title: Keeping Active in Residential Elderly
Acronym: KARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: HUR Labs (Unknown); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERN_16-1438
Record Dates: First submitted 2017-04-21; First posted 2017-05-05 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Frail Elderly Syndrome; Frailty; Physical Activity
Keywords: Frailty; Physical Activity; Resistance training
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention (Experimental): HUR resistance training intervention
  Interventions: Other: HUR equipment resistance training intervention
- Regular care (No Intervention): (Wait-list control)

INTERVENTIONS:
Other: HUR equipment resistance training intervention — Resistance training intervention
  Arms: Physical Activity Intervention

SUMMARY:
This trial will take the form of a feasibility study; designed to assess the feasibility of a proposed future clinical trial in this setting. This proposed future clinical trial is proposed to assess the impact of physical activity, in the form of specialised chair based physical activity intervention, on the physiological, psychological, cognitive, social and emotional health, and functional capacity of geriatric populations with pre-existing frailty within a residential care setting; recognising health as a holistic concept incorporating a multitude of inter-related dimensions. This feasibility study is single-centre (taking place at the Olivet Christadelphian care home, 17 Sherbourne Road, Acocks Green, Birmingham, United Kingdom ).

ELIGIBILITY:
Inclusion Criteria:

* Residents within the Olivet Christadelphian care home, 17 Sherbourne Road, Acocks Green, Birmingham, United Kingdom
* ≥ 65 years of age
* Frail according to the Fried Frailty criteria: meeting at least three of the five characteristics of frailty (Fried et al. 2001)
* Have the capacity to speak and read in English

Exclusion Criteria:

* Currently taking part in any other clinical trial which could potentially have an impact upon or influences the findings of the current study
* Currently terminally ill with life expectancy which is less than the duration of the follow-up of the study
* Severe sensory impairment which would profoundly impact on their capacity to undergo the interventions, even once appropriate adaptations have been made.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Feasibility assessments will occur post-intervention (six-weeks) and during the follow-up (12-weeks), assessing the feasibility of the study from baseline to follow up (12 weeks)
  The primary dependent variables of this feasibility study will relate to the eight primary areas of focus of feasibility studies (Bowen et al. 2009), relating to:
  * Acceptability
  * Demand
  * Implementation
  * Practicality
  * Adaptation
  * Integration
  * Expansion and
  * Limited-efficacy testing
  These eight aforementioned areas (all constituting the one variable of feasibility) will serve as the primary dependent variable for this study, in order to establish the feasibility of the proposed future clinical trial within this setting. The dependent variable of feasibility will be assessed through semi-structured interviews with study participants post intervention, while focus groups will be utilised with both the intervention implementers and study support staff in order to assess the primary dependent variable of the study.

SECONDARY OUTCOMES:
Cortisol (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Dehydroepiandrosterone-sulphate (DHEAS) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Serum cortisol: DHEAS ratio (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
C-Reactive proteins (CRP) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Inflammatory cytokine: Interleukin 6 (IL-6) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Inflammatory cytokine: Tumor Necrosis Factor alpha (TNFα) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Inflammatory cytokine: Interferon gamma (IFNy) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Handgrip strenght (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Leg Strength (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Leg power output (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Short Physical Performance Battery (SPPB) (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Katz Index of Independence in Activities of Daily Living (Katz ADL) (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Fried Frailty Phenotype (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Geriatric Depression Scale (GDS) (Psychological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Hospital Anxiety Depression Scale (HADS) (Psychological Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Psychological Dependent Variable: Perceived Stress Scale (PSS) (Psychological Dependent Variable | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
Standardized Mini-Mental State Examination (SMMSE) (Cognitive Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)
  Standardized Mini-Mental State Examination (SMMSE)
Interpersonal Support Evaluation List (Social Dependent Variable) | Pre-intervention (baseline), and post-intervention (six-weeks), follow-up (12-weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Anna Whittaker, Principal Investigator — University of Birmingham
Locations (1):
- Olivet Christadelphian care home, 17 Sherbourne Road, Acocks Green, Birmingham, United Kingdom, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Derived] Swales B, Ryde GC, Whittaker AC. A Mixed Methods Feasibility Study of Machine-Based Resistance Training With Prefrail Older Adults in Residential Care: The Keeping Active in Residential Elderly Trial II. J Aging Phys Act. 2024 Jan 23;32(2):244-263. doi: 10.1123/japa.2022-0170. Print 2024 Apr 1. PMID 38262397
- [Derived] Swales B, Ryde GC, Fletcher I, Whittaker AC. The reliability and suitability of strength assessments in frail and pre-frail older adults: recommendations for strength testing in older populations. BMC Geriatr. 2023 Dec 8;23(1):820. doi: 10.1186/s12877-023-04552-3. PMID 38066459
- [Derived] Swales B, Ryde GC, Whittaker AC. A Randomized Controlled Feasibility Trial Evaluating a Resistance Training Intervention With Frail Older Adults in Residential Care: The Keeping Active in Residential Elderly Trial. J Aging Phys Act. 2022 Jun 1;30(3):364-388. doi: 10.1123/japa.2021-0130. Epub 2021 Sep 11. PMID 34510020
- [Derived] Doody P, Lord JM, Whittaker AC. Assessing the feasibility and impact of an adapted resistance training intervention, aimed at improving the multi-dimensional health and functional capacity of frail older adults in residential care settings: protocol for a feasibility study. Pilot Feasibility Stud. 2019 Jul 5;5:86. doi: 10.1186/s40814-019-0470-1. eCollection 2019. PMID 31321070
- See also: Physical Activity and Nutritional INfluences In ageing (PANINI) project website — http://www.birmingham.ac.uk/generic/panini/index.aspx
- See also: Physical Activity and Nutritional INfluences In ageing (PANINI) project twitter — https://twitter.com/PANINI_EU